CLINICAL TRIAL: NCT00932035
Title: Reducing Extremity Lymphedema Through Axillary Lymphatic Preservation Surgery
Brief Title: Axillary Lymph Node Preservation Surgery in Reducing Lymphedema in Patients With Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Loss of principal investigator
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 11130
Record Dates: First submitted 2009-06-29; First posted 2009-07-02 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: breast cancer; axillary mapping; lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (reverse mapping guided axillary lymph node dissection) (Experimental): Patients receive isosulfan blue dye SC and then undergo reverse mapping-guided axillary lymph node dissection.
  Interventions: Procedure: axillary lymph node dissection; Drug: isosulfan blue based lymphatic mapping; Procedure: quality-of-life assessment; Other: Questionnaire administration
- Arm II (control) (Active Comparator): Patients undergo standard axillary lymph node dissection and then receive isosulfan blue dye SC.
  Interventions: Drug: isosulfan blue based lymphatic mapping; Procedure: axillary lymph node dissection; Procedure: quality-of-life assessment; Other: Questionnaire administration

INTERVENTIONS:
Procedure: axillary lymph node dissection — Undergo reverse mapping-guided axillary lymph node dissection
  Other Names: isosulfan blue dye; Lymphazurin blue dye
  Arms: Arm I (reverse mapping guided axillary lymph node dissection)
Drug: isosulfan blue based lymphatic mapping
  Other Names: isosulfan blue dye; Lymphazurin blue dye
Procedure: axillary lymph node dissection — Undergo standard axillary lymph node dissection
  Other Names: isosulfan blue dye; Lymphazurin blue dye
  Arms: Arm II (control)
Procedure: quality-of-life assessment — Ancillary studies
Other: Questionnaire administration — Ancillary studies

SUMMARY:
This pilot phase I and randomized phase II trial studies the best way to perform axillary lymph node preservation surgery and to see how well it works in preventing lymphedema in patients with breast cancer. Lymph node mapping may help in planning surgery to remove breast cancer and affected lymph nodes. It is not yet known whether reverse mapping guided axillary lymph node dissection is more effective than standard axillary lymph node dissection in preventing lymphedema.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To produce a map of the lymphatic drainage of the upper extremity as it relates to breast drainage, to determine the proportion of women undergoing axillary lymphadenectomy at risk for lymphedema. II. To determine if blue lymphatics contain lymph node metastases. III. To evaluate the incidence of lymphedema and associated other surgical related quality of life in those undergoing this procedure as compared to the current standard of care.

OUTLINE: This is a phase I study followed by a randomized phase II study.

PILOT PORTION: Patients receive isosulfan blue dye subcutaneously (SC) and then undergo reverse mapping-guided axillary lymph node dissection.

RANDOMIZED PORTION: Patients are randomized to 1 of 2 treatment arms. ARM I: Patients receive isosulfan blue dye subcutaneously (SC) and then undergo reverse mapping-guided axillary lymph node dissection. ARM II: Patients undergo standard axillary lymph node dissection and then receive isosulfan blue dye SC.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

- Patients diagnosed with breast cancer with a planned axillary lymph node dissection planned for breast cancer

Exclusion Criteria:

* Prior lymphedema in either arm
* Prior history of axillary surgery (except for sentinel node biopsies)
* Prior history of chest/axillary radiation
* Need for bilateral axillary node dissection surgery
* Prior neurologic deficits (either motor or sensory) in ipsilateral arm
* Known allergy to vital blue dyes
* No prior diagnosis of inflammatory breast cancer
* Cannot be pregnant or planning to continue breast-feeding immediately after surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Chen, MD, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - University of California, Davis Medical Center, Sacramento, California
  - University of North Carolina, Chapel Hill, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Reverse Mapping Guided Axillary Lymph Node Dissection): Patients receive isosulfan blue dye SC and then undergo reverse mapping-guided axillary lymph node dissection.
  axillary lymph node dissection: Undergo reverse mapping-guided axillary lymph node dissection
  isosulfan blue based lymphatic mapping
  quality-of-life assessment: Ancillary studies
- Arm II (Control): Patients undergo standard axillary lymph node dissection and then receive isosulfan blue dye SC.
  isosulfan blue based lymphatic mapping
  axillary lymph node dissection: Undergo standard axillary lymph node dissection
  quality-of-life assessment: Ancillary studies
  Questionnaire administration: Ancillary studies
Period: Overall Study
Arm/Group | Arm I (Reverse Mapping Guided Axillary Lymph Node Dissection) | Arm II (Control)
Started | 18 | 21
Completed | 18 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Reverse Mapping Guided Axillary Lymph Node Dissection) | Arm II (Control) | Total
Number analyzed (Participants) | 18 | 21 | 39
Age, Continuous [Median (Full Range); unit: years] | 52 [28 to 81] | 47 [32 to 73] | 50 [28 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 21 | 39

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Arm Lymphatics Above, at, or Below the Axillary Vein
Description: A Fisher's exact test with a one-sided alpha of 0.05 will be used to determine if the percentage of patients with arm lymphatics above, around, or below the axillary vein in the standard dissection group is superior to the experimental dissection group.
Time Frame: Up to 4 years
Population: Because of early termination the study did not accrue the planned number of subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Reverse Mapping Guided Axillary Lymph Node Dissection) | Arm II (Control)
Number analyzed (Participants) | 11 | 14
Participants
  Blue Lymphatic Channels Seen | 9 | 10
  Blue Lymphatic Channels Not Seen | 2 | 4
Statistical Analysis 1: Comparison: Arm I (Reverse Mapping Guided Axillary Lymph Node Dissection) vs Arm II (Control); Test type: Superiority — To achieve a power of 0.84, a sample size of 72 patients, evenly distributed is required. With 36 patients per group, a Fisher's exact test with a one-sided alpha of 0.05 will have a 84% power to detect the difference between the experimental group (axillary reverse mapping) of 5% or less and a control group (standard dissection) of 30% or more. Response estimates were chosen based on reported lymphedema rates; p = 0.45, Fisher Exact

2. Primary Outcome: Percentage of Patients With Positive Axillary Reverse Mapping (ARM) Identified Nodes
Description: A Fisher's exact test with a one-sided alpha of 0.05 will be used to determine if the percentage of patients with positive ARM identified nodes excised in the standard dissection group is superior to the experimental dissection group.
Time Frame: Up to 4 years
Population: Because of early termination the study did not accrue the planned number of subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Reverse Mapping Guided Axillary Lymph Node Dissection) | Arm II (Control)
Number analyzed (Participants) | 11 | 14
Participants
  Blue Lymph Nodes Seen | 4 | 4
  Blue Lymph Nodes Not Seen | 7 | 10
Statistical Analysis 1: Comparison: Arm I (Reverse Mapping Guided Axillary Lymph Node Dissection) vs Arm II (Control); Test type: Superiority; p = 0.50, Fisher Exact

3. Primary Outcome: Percentage of Patients With Lymphedema
Description: Difference between arms in patients developing lymphedema at any point during the study will be evaluated using chi-squared tests.
Time Frame: Up to 4 years
Population: Because of early termination the study did not accrue the planned number of subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Reverse Mapping Guided Axillary Lymph Node Dissection) | Arm II (Control)
Number analyzed (Participants) | 18 | 20
Participants
  Lymphedema Present | 4 | 6
  Lymphedema Not Present | 14 | 14
Statistical Analysis 1: Comparison: Arm I (Reverse Mapping Guided Axillary Lymph Node Dissection) vs Arm II (Control); Test type: Superiority; p = 0.59, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 28 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Groups:
- Arm I (Reverse Mapping Guided Axillary Lymph Node Dissection): Patients receive isosulfan blue dye SC and then undergo reverse mapping-guided axillary lymph node dissection.
  axillary lymph node dissection: Undergo reverse mapping-guided axillary lymph node dissection
  isosulfan blue based lymphatic mapping
  quality-of-life assessment: Ancillary studies
  Questionnaire administration: Ancillary studies
Arm/Group | Arm I (Reverse Mapping Guided Axillary Lymph Node Dissection) | Arm II (Control)
Serious Adverse Events (participants affected / at risk) | 1/18 | 1/21
Other Adverse Events (participants affected / at risk) | 13/18 | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Reverse Mapping Guided Axillary Lymph Node Dissection) (N=18) | Arm II (Control) (N=21)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Reverse Mapping Guided Axillary Lymph Node Dissection) (N=18) | Arm II (Control) (N=21)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 2 (2) | 0 (0)
Localized edema (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (3) | 2 (4)
Breast infection (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 2 (2) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
JP Drain Blood Leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Left Shoulder Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pain-post op (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast Swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated early due to loss of principal investigator. As a result accrual of subjects and data collection are incomplete.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes